CLINICAL TRIAL: NCT06949943
Title: Enhancing Quality of Patient Experience Via an Innovative Reduction of Pre-Operative Anxiety
Brief Title: Pre-Operative Guided Meditation to Reduce Pre-Operative Anxiety in Patients Undergoing Cancer-Directed Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Maryanna Klatt, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OSU-24146; NCI-2025-01389 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2025-03-25; First posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Hematopoietic and Lymphatic System Neoplasm; Malignant Solid Neoplasm
MeSH Terms: interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (guided meditation) (Experimental): Patients listen to 10 minutes of guided meditation prior to surgery.
  Interventions: Behavioral: Behavioral Intervention; Other: Electronic Health Record Review; Other: Survey Administration
- Arm II (noise cancelling headphones) (Active Comparator): Patients wear noise cancelling headphones for 10 minutes prior to surgery.
  Interventions: Behavioral: Behavioral Intervention; Other: Electronic Health Record Review; Other: Survey Administration

INTERVENTIONS:
Behavioral: Behavioral Intervention — Listen to guided meditation
  Other Names: Behavior Conditioning Therapy; Behavior Modification; Behavior or Life Style Modifications; Behavior Therapy; Behavioral Interventions; Behavioral Modification; Behavioral Therapy; Behavioral Treatment; Behavioral Treatments
  Arms: Arm I (guided meditation)
Behavioral: Behavioral Intervention — Wear noise cancelling headphones
  Other Names: Behavior Conditioning Therapy; Behavior Modification; Behavior or Life Style Modifications; Behavior Therapy; Behavioral Interventions; Behavioral Modification; Behavioral Therapy; Behavioral Treatment; Behavioral Treatments
  Arms: Arm II (noise cancelling headphones)
Other: Electronic Health Record Review — Ancillary studies
Other: Survey Administration — Ancillary studies

SUMMARY:
This clinical trial tests how well guided meditation, compared to silence, works to reduce pre-operative anxiety in patients undergoing cancer-directed surgery. Pre-operative anxiety affects patient experience and has been found to be a predictor of severe post-operative pain and chronic pain after surgery, influencing the success and quality of a patient's recovery. While medication is often prescribed to improve anxiety symptoms, research has showed that mindfulness techniques can be used to decrease anxiety, improve comfort, and can impact both psychological and physiologic symptoms. Completing pre-operative guided meditation may work well to reduce pre-operative anxiety in patients undergoing cancer directive surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To improve is pre-operative patient anxiety in surgical settings.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients listen to 10 minutes of guided meditation prior to surgery.

ARM II: Patients wear noise cancelling headphones for 10 minutes prior to surgery.

After completion of study intervention, patients are followed up for up to 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be recruited among patients who are scheduled for cancer-directed surgery
* Participants must be 18 years or older

Exclusion Criteria:

* Participants will be excluded from the study if they cannot speak English (as the meditation is recorded in English)
* Currently incarcerated
* Have a diagnosis of dementia
* Are admitted to the intensive care unit (ICU)
* Have a hearing impairment that would make them unable to hear the recorded meditation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-03-14 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Pre-operative anxiety (PROMIS Anxiety scale) | Pre and post intervention, approximately 10 minutes
  Measured with the Patient Reported Outcome Measurement Information System Anxiety. PROMIS Anxiety short form is an 8-item scale used to assess anxiety in individuals 18 years or older. Each item is on a 5-point scale to be summed, with higher scores indicating greater anxiety.
Pre-operative anxiety (single-item visual analog scale) | Pre and post intervention, approximately 10 minutes
  Measured by a single-item visual analog scale. The single-item visual analog scale will be used to assess momentary anxiety. The item will ask, "On a scale of 1 to 10, how anxious do you feel right now?" and patients will rate the level of anxiety on a scale of 0 to 10 (0=not at all anxious, 10=extremely anxious).

SECONDARY OUTCOMES:
Post-operative opiate use | Up to 6 months post intervention
  Will be extracted from the electronic medical record via chart review. Days of opioid use will be calculated and compared between intervention and control groups.
Post-operative morphine equivalent dose | Up to 6 months post intervention
  Will be extracted from the electronic medical record via chart review. Daily morphine equivalent dose for each opioid prescribed will be calculated and compared between intervention and control groups.
Post-operative average daily morphine | Up to 6 months post intervention
  Will be extracted from the electronic medical record via chart review. Average daily morphine equivalent dose will be calculated and compared between intervention and control groups.
Length of stay | Up to 6 months post intervention
  Will be extracted from the electronic medical record via chart review.

CONTACTS AND LOCATIONS:
Overall Officials: Maryanna Klatt, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu